CLINICAL TRIAL: NCT01586767
Title: A Phase II Study of Intensity-Modulated or Proton Radiation Therapy for Locally Advanced Sinonasal Malignancy
Brief Title: Intensity-Modulated or Proton Radiation Therapy for Sinonasal Malignancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Annie W. Chan, MD, Assistant Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-308; 2P01CA021239-29 (NIH)
Record Dates: First submitted 2011-10-21; First posted 2012-04-27 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Adenoid Cystic Carcinoma; Squamous Cell Carcinoma; Sinonasal Carcinoma; Sinonasal Undifferentiated Carcinoma; Mucoepidermoid Carcinoma; Schneiderian Carcinoma; Myoepithelial Carcinoma; Esthesioneuroblastoma; Melanoma
Keywords: Nasal cavity; Salivary gland tumors; Hard palate; Sinus; Soft Palate; Lacrimal Apparatus
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Carcinoma, Squamous Cell; Sinonasal undifferentiated carcinoma; Carcinoma, Mucoepidermoid; Esthesioneuroblastoma, Olfactory; Melanoma; Fistula | interventions — Protons; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton beam therapy (Active Comparator): Subjects treated at Massachusetts General Hospital with proton beam therapy
  Interventions: Radiation: Proton radiation therapy
- IMRT (Active Comparator): Intensity-modulated radiation therapy at institutions other than Massachusetts General Hospital
  Interventions: Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Radiation: Proton radiation therapy — Daily proton radiation therapy
  Arms: Proton beam therapy
Radiation: Intensity-modulated radiotherapy — Daily intensity-modulated radiotherapy
  Other Names: IMRT
  Arms: IMRT

SUMMARY:
The purpose of this study is to test the hypothesis that 1)intensity-modulated radiotherapy (IMRT) or proton radiation therapy would result in improved local control rate and lowered toxicity compared to conventional radiotherapy, and 2) proton radiation therapy would result in equivalent or improved local control rate with similar or lower toxicity compared to IMRT, in the treatment of locally advanced sinonasal malignancy.

Data from retrospective studies suggest that IMRT or proton radiation therapy resulted in promising outcome in patients with sinonasal malignancy. To this date, no prospective study has been conducted to evaluate the outcome of sinonasal cancer treated with IMRT or proton radiation therapy. This Phase II trial is the first prospective study conducted to determine the treatment outcome and toxicity of IMRT or proton in the treatment of sinonasal cancer.

IMRT and proton radiation therapy are the two most established and most commonly employed advanced radiotherapy techniques for the treatment of sinonasal cancer. It is highly controversial whether one is superior to the other in terms of local control and toxicity outcome. It is also not clear if a subset of patients would benefit more from one treatment technology versus the other.

Due to the rarity and heterogeneity of sinonasal malignancies and the fact that proton beam is only available at a few centers in the United States, it is not feasible at present to do a Phase III study randomizing patients between IMRT and proton radiation therapy. In this study, a planned secondary analysis will be performed, comparing the treatment and toxicity outcome between IMRT and proton. The data on the IMRT and proton comparison from this trial will be used to design future multi-center prospective trials and to determine if randomized trial is necessary.

In this study, the treatment technique employed for an individual case will not be determined by the treating physician(s), but rather by the most advanced technology available at the treating institution for the treatment of the sinonasal cancer. At the Massachusetts General Hospital (MGH), proton beam therapy will be used for patients who meet the eligibility criteria. For institutions where protons are not available or institutions where the proton planning systems have not been optimized, IMRT exclusively will be used for the treatment of sinonasal cancer. Patient and tumor characteristics are expected to be comparable between IMRT- and proton- institutions

DETAILED DESCRIPTION:
Subjects will receive daily proton radiation treatment as outpatients at the Francis H. Burr Proton Center at Massachusetts General Hospital. The subjects may also receive concurrent standard chemotherapy every week during their radiation therapy. This chemotherapy is considered standard treatment for their cancer and is not being done for research purposes.

In addition to daily radiation treatments, subjects will have the following tests every week: review of side effects; physical exam, including weight, height, neurological exam and vital signs; and blood tests, only for those subjects also receiving chemotherapy.

Subjects will be followed for 5 years after the completion of study treatment. The first follow-up visit will be 6-8 weeks after completion of study treatment. Additional follow-up visits will be performed every 3 months during the first 2 years following completion of radiation then every 6 month during years 3-5. At each follow-up visit, subjects will receive a physical exam, chest CT scan (at 1st follow-up visit then at least every 6 months), a CT or MRI tumor assessment (at 1st follow-up visit then at least every 6 months), quality-of-life questionnaire, hearing test, neuro-ophthalmology test, and neurocognitive test.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven, within 16 weeks prior to study entry, sinonasal adenoid cystic carcinoma, adenocarcinoma, mucoepidermoid carcinoma, squamous cell carcinoma, including sinonasal carcinoma, sinonasal undifferentiated carcinoma, Schneiderian carcinoma, myoepithelial carcinoma, undifferentiated carcinoma, esthesioneuroblastoma, or melanoma AJCC 7th edition Stage III - IVA/B tumors, or with skull base or intracranial extension. Pathology must be confirmed by review at the treating institution.
* Patients with biopsy proven locally advanced sinus, nasal cavity, hard palate, soft palate, major or minor salivary gland tumors, or lacrimal apparatus, with nasal cavity, sinus, auditory canal, or skull base involvement are eligible.
* Eastern cooperative oncology group (ECOG) performance status 0 - 1 or Karnofsky Performance Status ≥ 70. (Appendix B)
* All patients must undergo pre-treatment evaluation of tumor extent prior to study entry through imaging studies and clinical examinations, including CT and/or MRI of skull base, brain and neck within 28 days prior to study entry; physical examination +/- nasal endoscopy within 28 days prior to study entry; and CT of the chest within 60 days prior to study entry.
* Nutritional and general physical condition must be considered compatible with the proposed radiation +/- chemotherapy treatment.
* Normal organ and marrow function

Exclusion Criteria:

* Active alcohol addiction
* Pregnant or breastfeeding
* Receiving any other study agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin for subjects who will receive chemotherapy
* Evidence of distant metastases or distant leptomeningeal metastases
* Previous irradiation for head and neck tumor, skull base, or brain tumors
* Uncontrolled intercurrent illness
* History of a different malignancy unless disease-free for at least 2 years and are deemed by the investigator to be at low-risk for recurrence. Individuals with the following cancers are eligible if diagnosed and treated for cure within the past 2 years: cervical cancer in situ, carcinoma in situ of the breast, and basal cell or squamous ceel carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-07-12 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Local Control Rates | 2 years
  To determine the local control rates with IMRT or proton radiation therapy at 2 years.

SECONDARY OUTCOMES:
Vision preservation | 5 years
  To determine the late visual-orbital late effects of IMRT or proton beam
Regional control | 2 years
  To determine the regional control at 2 years after IMRT or proton
Survival | 5 years
  To determine the long-term survival at 5 years after IMRT or proton
QOL | 5 years
  To assess quality-of-life (QOL) outcomes after IMRT or proton
Patterns of Tumor Relapse | 5 years
  To determine the patterns of tumor relapse after IMRT or proton
Local control | 5 years
  To determine long-term local control after IMRT or proton
Neurocognitive function | 5 years
  To determine long-term neurocognitive function after IMRT or proton

CONTACTS AND LOCATIONS:
Overall Officials: Annie W Chan, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota